CLINICAL TRIAL: NCT03478189
Title: The Added Value of Intraoperative CT Scanner and Screw Navigation in Operative Treatment of Displaced Acetabular Fracture With Dome Impaction
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: OARM impactionTOIT
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Acetabular Fracture; Acetabular Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: use of O-arm surgical imaging — during acetabular fracture surgery , use of O-arm surgical imaging with

SUMMARY:
The acetabulum fracture result from a trauma with high energy at the young adult or from a trauma of low energy at the old osteoporotic patient. Anatomic reduction is known to be necessary to give functional result to patient.However, it's technically difficult because of the pelvic bone conformation.

The presence of dome impaction makes the surgery more difficult. Per operatory scanner associated to 3D navigation is proved his value-added in spinal surgery.The aim of the study is show that this association permit a technical improvement for the surgeon in the precision of fracture reduction.and restore the articular congruence.

ELIGIBILITY:
Inclusion Criteria:

* age> 18
* surgery for acetabular fracture within 30 days
* with dome impaction

Exclusion Criteria:

* disability of inferior limb

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient hospitalized in GHPSJ from april 2016 and october 2017
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
dome impaction reduction measurement | day1
  dome impaction reduction measurement on scanner per operatory and post operatory

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume RIOUALLON, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France